CLINICAL TRIAL: NCT03367559
Title: An Open Label Study to Evaluate Immunogenicity, Safety, and Reactogenicity of Rotavac® (Live Attenuated Rotavirus Vaccine) as a 3-dose Series in Healthy Infants Aged Between 6 Weeks and 8 Weeks in Vietnam
Brief Title: Evaluate Immunogenicity, Safety, and Reactogenicity of Rotavac® in Healthy Infants Aged Between 6-8 Weeks in Vietnam
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Institute of Clinical Research and Clinical Trial Support for Vaccine and Biological Products (Other)
Collaborators: Bharat Biotech International Limited (Industry)
Responsible Party: Principal Investigator, Pham Ngoc Hung, MD PhD Assoc, Principal Investigator, Vietnam Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VX-2017.01
Record Dates: First submitted 2017-12-05; First posted 2017-12-08 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Rotavirus Infections
Keywords: Rotavirus; ROTAVAC; Vaccine; Vietnam
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Masking Description: An open label study to evaluate immunogenicity, safety, and reactogenicity of Rotavac® (live attenuated rotavirus vaccine) as a 3-dose series in healthy infants aged between 6 weeks and 8 weeks in Vietnam
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rotavirus Vaccine (Experimental): 3 dose, interval for each dose is 4 weeks. The first dose will be received at 6-8 weeks of age.
  Interventions: Biological: ROTAVAC®

INTERVENTIONS:
Biological: ROTAVAC® — Rotavac® is in frozen form and is thawed till fully liquid prior to administration.

SUMMARY:
An open label study to evaluate immunogenicity, safety, and reactogenicity of Rotavac® (live attenuated oral rotavirus vaccine) as a 3-dose series in healthy infants aged between 6 weeks and 8 weeks in Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants as established by medical history and clinical examination before entering the study.
* Age: 6-8 weeks
* Weight ≥ 2.5kg at birth.
* Infants received EPI vaccines at birth (i.e., OPV, BCG and/or Hep B)
* Parental ability and willingness to provide informed consent.
* Parent who intends to remain in the area with the participant during the study period.

Exclusion Criteria:

* Presence of diarrhea or vomiting in the previous 72 hours or on the day of enrollment (temporary exclusion).
* Presence of fever (temperature ≥37.5oC) or hypothermia (temperature ≤35.5oC) on the day of enrollment (temporary exclusion).
* Concurrent participation in another clinical trial.
* Presence of significant malnutrition or any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, immunological, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination which would compromise the infant's health or is likely to result in non-conformance to the protocol.
* History of congenital abdominal disorders, intussusception, abdominal surgery
* Known or suspected impairment of immunological function based on medical history and physical examination.
* Prior receipt of rotavirus vaccine.
* A known sensitivity or allergy to any components of the study medication.
* Major congenital or genetic defect.
* Participant's parents not able, available or willing to accept active follow-up by the study staff.
* Has received any immunoglobulin therapy and/or blood products since birth or planned administration during the study period.
* History of chronic administration (defined as more than 14 days) of immunosuppressants including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study.
* History of any neurologic disorders or seizures.
* Any medical condition in the parents/infants that, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parent's/legally acceptable representative's ability to give informed consent.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Frequency and rate of the AEs within 30 minutes after vaccination | 30 minutes after vaccination
  Frequency and rate of the adverse effects and severity of immediate adverse events (Local and General) within 30 minutes after vaccination
Frequency and rate of the AEs within 7 days after vaccination | for 7 days after each vaccination
  Frequency and rate of adverse effects and severity of solicited adverse events (Local and General) within 7 days after each vaccination
Frequency and rate of the AEs during 28 days after vaccination | for 28 days after vaccination
  Frequency and rate of adverse effects and severity of unsolicited adverse events (Local and General) during 28 days after each vaccination
Frequency and rate of the SAEs during 28 days after vaccination | for 28 days after vaccination
  Frequency and rate of adverse effects and severity of Serious Adverse Events (Local and General) during 28 days after each vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Thai Binh Health Center, Thái Bình, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided